CLINICAL TRIAL: NCT04594603
Title: Changes of Macular Vasculature After Uncomplicated Phacoemulsification Surgery Using Optical Coherence Tomography Angiography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dina Tadros, Lecturer of Ophthalmology, Tanta University, Egypt, Tanta University
Other Study IDs: 34082/9/20
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Phacoemulsification

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group(1): Cataract with no diabetic retinopathy
  Interventions: Other: Phacoemulsification for cataract
- Group (2): Cataract associated with diabetic retinopathy
  Interventions: Other: Phacoemulsification for cataract

INTERVENTIONS:
Other: Phacoemulsification for cataract — Phacoemulsification for removal of cataract

SUMMARY:
To record the vascular changes that may be present in the macular after uncomplicated phacoemulsification surgery by using OCTA, a comparative study between healthy and diabetic patients

DETAILED DESCRIPTION:
A prospective study of 30 patients with senile or complicated cataract scheduled to do phacoemulsification surgery in Tanta University Hospital

Two groups will be divided:

1. Group (1): Cataract will no diabetic retinopathy
2. Group (2): Cataract associated with diabetic retinopathy.

All patients will be subject to Full ophthalmologic examination before the surgery. Imaging will include OCTA. OCTA will be performed using cirrus OCT (Zeiss, Inc., USA). High-quality 6 x 6 mm OCTA macular scans and 3 × 3-mm papillary scan with strong signal-noise ratio with adequate centration on the fovea and optic nerve head respectively will be selected.

Segmentation will be used to evaluate superﬁcial and deep capillary retinal plexus projections in addition to the choriocapillaries. If errors in segmentation were detected, manual correction would be performed. The superﬁcial retinal capillary plexus (SCP) will be delineated with an inner boundary at the internal limiting membrane (ILM) and an outer boundary 10 µm inside the inner plexiform layer (IPL). The deep retinal capillary plexus (DCP) will be segmented with an inner boundary 10 µm inside the IPL and an outer boundary at 10 µm beneath the outer plexiform layer (OPL).

The vessel density metric from enface OCT angiogram will be used as an indicator of macular retinal and papillary perfusion. Vessel density (VD) analysis computes the percentage of area occupied by OCTA detected vasculature in a measured area. Choriocapillaries flow voids will be computed to assess choriocapillaries circulation.

The measurements of the OCTA, axial length, intraocular pressure will be obtained before the phacoemulsification surgery. Optical coherence tomography and IOP measurements will also be obtained 1 week after surgery.

ELIGIBILITY:
Inclusion Criteria:

* - Presence of a nuclear, cortical cataract or complicated cataract due to diabetic mellitus
* Intraocular pressure (IOP) of 21 mm Hg or lower
* Axial length (AL) between 20.0 mm and 25.0 mm.

Exclusion Criteria:

* Eyes with an AL longer than 25.0 mm or shorter than 20.0 mm,

  * IOP higher than 21 mm Hg,
  * History of ocular trauma or intraocular surgery, or any abnormal intraocular findings
  * Poor OCT-A images because of severe cataracts or unstable fixation
  * Any signs of intraoperative or postoperative complications

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a prospective study of 30 patients with senile or complicated cataract scheduled to do phacoemulsification surgery in Tanta University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
To record the vascular changes that may be present in the macular after uncomplicated phacoemulsification surgery by using OCTA | 1 week after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospital, Tanta, El-Garbeia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 3 months
Access Criteria: Link

REFERENCES:
- [Result] Mirshahi A, Hohn F, Lorenz K, Hattenbach LO. Incidence of posterior vitreous detachment after cataract surgery. J Cataract Refract Surg. 2009 Jun;35(6):987-91. doi: 10.1016/j.jcrs.2009.02.016. PMID 19465281
- [Result] Ripandelli G, Coppe AM, Parisi V, Olzi D, Scassa C, Chiaravalloti A, Stirpe M. Posterior vitreous detachment and retinal detachment after cataract surgery. Ophthalmology. 2007 Apr;114(4):692-7. doi: 10.1016/j.ophtha.2006.08.045. Epub 2007 Jan 17. PMID 17208303
- [Result] Rossetti L, Autelitano A. Cystoid macular edema following cataract surgery. Curr Opin Ophthalmol. 2000 Feb;11(1):65-72. doi: 10.1097/00055735-200002000-00010. PMID 10724830
- [Result] Flach AJ. The incidence, pathogenesis and treatment of cystoid macular edema following cataract surgery. Trans Am Ophthalmol Soc. 1998;96:557-634. No abstract available. PMID 10360304
- [Result] Kim SJ, Equi R, Bressler NM. Analysis of macular edema after cataract surgery in patients with diabetes using optical coherence tomography. Ophthalmology. 2007 May;114(5):881-9. doi: 10.1016/j.ophtha.2006.08.053. Epub 2007 Feb 1. PMID 17275910
- [Result] Or C, Sabrosa AS, Sorour O, Arya M, Waheed N. Use of OCTA, FA, and Ultra-Widefield Imaging in Quantifying Retinal Ischemia: A Review. Asia Pac J Ophthalmol (Phila). 2018 Jan-Feb;7(1):46-51. doi: 10.22608/APO.201812. Epub 2018 Feb 13. PMID 29436208
- [Result] Sorour OA, Sabrosa AS, Yasin Alibhai A, Arya M, Ishibazawa A, Witkin AJ, Baumal CR, Duker JS, Waheed NK. Optical coherence tomography angiography analysis of macular vessel density before and after anti-VEGF therapy in eyes with diabetic retinopathy. Int Ophthalmol. 2019 Oct;39(10):2361-2371. doi: 10.1007/s10792-019-01076-x. Epub 2019 May 22. PMID 31119505